CLINICAL TRIAL: NCT04051853
Title: Population Pharmacokinetics and Pharmacodynamics of Sorafenib in HCC Patients With Child-Pugh B Liver Cirrhosis (SORBE-trial)
Brief Title: Sorafenib PK in Patients With Advanced HCC and Child-Pugh B
Acronym: SORBE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Heinz-Josef Klumpen, Medical Oncologist & Principle Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014_078#B2014419a
Record Dates: First submitted 2016-02-11; First posted 2019-08-09 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: BCLC Stage C HCC; CP-B Liver Cirrhosis
Keywords: HCC; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sorafenib with midazolam clearance test (Experimental): Before start of treatment patients receive a single oral dose of midazolam to phenotype CYP3A4 activity. Blood samples will be taken at several time points to measure sorafenib and midazolam concentrations.
  Patients will receive sorafenib at a starting dose of 200 mg twice daily. In the absence of toxicity dosage will be escalated with weekly intervals up to 400 mg BID (max dose).
  Interventions: Drug: Sorafenib; Other: Midazolam clearance test
- Sorafenib with CYP cocktail test (Experimental): In this subgroup of 15 patients (in the Academic Medical Center Amsterdam), the midazolam test will be replaced by an oral cocktail of subclinical doses of caffeine, midazolam, omeprazole, warfarin and metoprolol and will be repeated after 4 weeks of treatment to assess the influence of sorafenib on cytochrome P450 (CYP) 1A2, 3A4, 2C19, 2C9 and 2D6 activity, respectively.
  Patients will receive sorafenib at a starting dose of 200 mg twice daily. In the absence of toxicity dosage will be escalated with weekly intervals up to 400 mg BID (max dose).
  Interventions: Drug: Sorafenib; Other: CYP cocktail clearance test

INTERVENTIONS:
Drug: Sorafenib — Patients will receive sorafenib at a starting dose of 200 mg twice daily. In the absence of toxicity dosage will be gradually escalated up to 400 mg BID.
Other: Midazolam clearance test — Before start of treatment patients receive a single oral dose of midazolam to phenotype CYP3A4 activity. Blood samples will be taken at several time points to measure sorafenib and midazolam concentrations.
  Arms: Sorafenib with midazolam clearance test
Other: CYP cocktail clearance test — In a subgroup of 15 patients (in the Academic Medical Center Amsterdam), this test will be replaced by an oral cocktail of subclinical doses of caffeine, midazolam, omeprazole, warfarin and metoprolol and will be repeated after 4 weeks of treatment to assess the influence of sorafenib on cytochrome P450 (CYP) 1A2, 3A4, 2C19, 2C9 and 2D6 activity, respectively.
  Arms: Sorafenib with CYP cocktail test

SUMMARY:
Sorafenib has proven efficacy in advanced hepatocellular carcinoma (HCC). Most patients with HCC have impaired liver function due to underlying liver cirrhosis. The severity of liver cirrhosis might have implications on sorafenib metabolism. To date, no data showing unequivocal activity and tolerability of sorafenib in patients with moderate cirrhosis (Child-Pugh (CP)-B) have been published.

To specifically address this issue, this study aims to explore population pharmacokinetics of sorafenib and to explore the relationship between sorafenib exposure and its efficacy and toxicity in CP-B patients with irresectable HCC.

DETAILED DESCRIPTION:
Study design:

This is a prospective, open-label, national, multicenter observational study to investigate the tolerability, pharmacokinetics and clinical activity of sorafenib and its metabolites in patients with HCC and CP-B liver cirrhosis

Study population:

45 Patients with BCLC stage C HCC and CP-B liver cirrhosis

Treatment:

All patients will receive sorafenib at a starting dose of 200 mg twice daily. In the absence of toxicity dosage will be gradually escalated up to 400 mg BID.

Before start of treatment patients receive a single oral dose of midazolam to phenotype CYP3A4 activity. Blood samples will be taken at several time points to measure sorafenib and midazolam concentrations.

In a subgroup of 15 patients (in the Academic Medical Center Amsterdam), this test will be replaced by an oral cocktail of subclinical doses of caffeine, midazolam, omeprazole, warfarin and metoprolol and will be repeated after 4 weeks of treatment to assess the influence of sorafenib on cytochrome P450 (CYP) 1A2, 3A4, 2C19, 2C9 and 2D6 activity, respectively.

Main study parameters/endpoints:

Primary

1. Exposure and intra- and inter-patient variability in exposure to sorafenib and its metabolites
2. Identification of predictive factors for sorafenib exposure, i.e. bilirubin, CYP3A4 activity Secondary
3. Correlation between sorafenib exposure and adverse events and progression free survival
4. Difference in exposure to 5 CYP probe drugs following administration of an oral cocktail of these agents after 4 weeks of sorafenib treatment in comparison with exposure to these cocktail probe drugs before initiation of sorafenib (substudy in 15 patients).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Enrolled patients will be admitted in the hospital for three 8h visits for pharmacokinetic (PK) sampling of sorafenib and midazolam or the drug cocktail (used for CYP phenotyping). All PK blood samples will be drawn via an intravenous catheter. The total amount of blood taken will be ca 70 ml. The risks of these procedures are low.

Patients with advanced HCC and (mild) CP-B liver cirrhosis are often considered poor candidates for sorafenib treatment due to decreased tolerability. The aim of this study is to look for treatment optimization strategies of sorafenib in this subgroup of advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Diagnosis of HCC: diagnosis based on the following criteria:

  1. 1 radiologic technique: Focal lesion >1 cm with arterial hypervascularization in 4-phase CT or dynamic contrast enhanced MRI OR
  2. 2 coincidental dynamic radiologic techniques (CT or MRI) in case one imaging technique is non-conclusive and lesion > 1 cm OR
  3. biopsy proven HCC
* Patients with advanced HCC - BCLC stage C
* Cancer related symptoms (symptomatic tumors, ECOG Performance status 1-2), macrovascular invasion (either segmental or portal invasion) or extrahepatic spread (lymph node involvement or distant metastases)
* Not eligible for TACE (; i.e. diffuse tumors, tumors larger than 5 cm)
* Not eligible for curative resection or RFA
* Patients with CP-B liver cirrhosis (CP-B score 7 or 8)
* Capable of giving written informed consent
* History of organ transplant (including prior liver transplantation) is allowed
* HIV, congenital immune defect, any immunosuppressive therapy for autoimmune disease (rheumatoid arthritis) is allowed

Exclusion Criteria:

Subjects will not be enrolled in the study if any of the following criteria apply:

* CP-B9 liver cirrhosis
* CP-C liver cirrhosis
* Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
* Concurrent antitumoral treatment for HCC or other malignancies
* Not eligible for sorafenib treatment
* Bilirubin > 51 micromol/L
* If female, pregnant or breast feeding (females of child-bearing potential must use adequate contraception and must have a negative pregnancy test performed within 7 days prior to inclusion into this study)
* If male, not using adequate birth control measures
* One or more of the following: - WBC <2,500 cells/mm3, - ANC <1,500 cells/mm3, - platelets <50,000/mm3,
* ECOG performance status >2
* Patients with known GFR <30 mL/min/1.73m2
* Significant cardiovascular disease; e.g., myocardial infarction within 6 months of inclusion, chronic heart failure (New York Heart Association class III or IV), unstable coronary artery disease
* Uncontrolled hypertension i.e. systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mm Hg despite optimal medical management (2 classes of antihypertensive drugs)
* History of hemorrhage / bleeding events of grade 3 or worse within 30 days before inclusion into this study
* Previous variceal bleeding within the past 3 months

Additional exclusion criteria for cocktail test

* Consumption of grapefruit or grapefruit juice and/or kumquats, pummelos, exotic citrus fruit (i.e., star fruit, bitter melon) or grapefruit hybrids from seven days prior to the first dose of cocktail.
* Use of herbal medicine or medication that induce or inhibit CYP3A4/5, CYP2C9, CYP2D6, CYP1A2 and CYP2C19
* Use of omeprazole, warfarin, metoprolol, caffeine or midazolam (=medication of the probe cocktail)
* Concurrent anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sorafenib exposure (AUC). | Through study completion, an average of 3 months
  Area under the plasma concentration versus time curve (AUC). Exposure and intra- and inter-patient variability in exposure to sorafenib. The population PK analysis will be performed using nonlinear mixed effects modelling (NONMEM). Predictive factors for sorafenib exposure, i.e. bilirubin, CYP3A4 activity, shall be explored.
Sorafenib peak plasma concentration | Through study completion, an average of 3 months
  Peak plasma concentration (Cmax) for sorafenib.
Sorafenib N-oxide exposure (AUC) | Through study completion, an average of 3 months
  Area under the plasma concentration versus time curve (AUC) for the main sorafenib metabolite (N-oxide sorafenib). Exposure and intra- and inter-patient variability in exposure to N-oxide sorafenib. The population PK analysis will be performed using nonlinear mixed effects modelling (NONMEM). Predictive factors for N-oxide sorafenib exposure, i.e. bilirubin, CYP3A4 activity, shall be explored.
Sorafenib N-oxide peak plasma concentration. | Through study completion, an average of 3 months
  Peak plasma concentration (Cmax) for the main sorafenib metabolite (N-oxide sorafenib).

SECONDARY OUTCOMES:
Adverse events according to CTCAE v4.0 | Through study completion, an average of 3 months.
  Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to sorafenib or drug cocktail. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded while receiving treatment and for 30 days after the last dose of Sorafenib, in order to detect delayed toxicity. Toxicity will be scored according NCI CTCAE version 4.0 The population PK analysis will be performed using nonlinear mixed effects modelling (NONMEM). Power calculations are not possible in NONMEM. Nevertheless, as a rule of thumb, 40 patients allow one to identify ca. 3 clinical significant correlations between PK parameters and patient characteristics. To be sure to have 40 evaluable patients we aim to recruit 45 patients.
Progression-free survival | Untill Progression or death (0-24 months)
  Progression free survival (PFS) is defined as the time from the date of start sorafenib to the first date of progressive disease (symptomatic or objective) or death to any cause, whichever occurs first.
Overall survival | Untill last follow-up or death (0-24 months)
  Overall surval is defined as the time from start sorafenib, to death or censored at last follow-up.
CYP activity | 4 weeks
  In order to assess CYP3A4 activity prior to the start of sorafenib treatment, a single oral dose of 0.03 mg/kg midazolam will be administered.
  Substudy in 15 patients: Difference in exposure to 5 CYP probe drugs following administration of an oral cocktail of these agents after 4 weeks of sorafenib treatment in comparison with exposure to these cocktail probe drugs before initiation of sorafenib.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Klümpen, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Ferry ALM Eskens, MD PhD, Principal Investigator — Erasmus MC Cancer Institute, Rotterdam; R. Bart Takkenberg, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Ron Mathot, PharmD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Hans Romijn, MD PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands